CLINICAL TRIAL: NCT03083223
Title: Comparison of Five Different Positions on Peripheral Oxygen Saturation and Vital Signs in Patients With Lung Disease
Brief Title: Positions and Peripheral Oxygen Saturation
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Leyla Khorshitd, Professor Dr., Ege University
Other Study IDs: 2013/44-19
Record Dates: First submitted 2017-03-06; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Lung Diseases
Keywords: patient positioning; lung diseases; oxygenation; hemodynamic parameters; vital signs
MeSH Terms: conditions — Lung Diseases | interventions — Patient Positioning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- lung disease: Patients with lung disease
  Interventions: Other: position

INTERVENTIONS:
Other: position — Subjects were placed consecutively in random order in five different positions. SaO2 and vital signs were measured at each position after 10, 25, and 40 minutes.

SUMMARY:
The subjects were placed consecutively in random order in the five different positions by drawing lots. Oxygen saturation (SaO2) and vital signs (pulse rate, respiratory rate, systolic blood pressure, diastolic blood pressure and body temperature) were measured in each position at 10, 25 and 40 minutes.

DETAILED DESCRIPTION:
The semi-seated position in bed at 45°: SSPB-45° The semi-seated position in bed at 60° :SSPB-60° Seated position in bed at 90°: SPB-90° Lying on the right side of the body at 45°: LRSB-45° , Lying on the left side of the body at 45°: LLSB-45°

A questionnaire which consisted of a Subjects' Introduction Form and a Vital Signs-SaO2 Record Form was used in collecting the data.

The subjects were placed consecutively in random order in the five different positions, SSPB-45°, SSPB-60°, SPB-90°, LRSB-45°, and LLSB-45°, by drawing lots. Oxygen saturation (SaO2) and vital signs (pulse rate, respiratory rate, systolic blood pressure, diastolic blood pressure and body temperature) were measured in each position at 10, 25 and 40 minutes. Oxygen saturation and vital signs were measured with a finger pulse oximeter (Nellcor N-560). Nail polish was removed before measurement of oxygen saturation, and if there was any physical restraint on subjects it was removed. Body temperature was measured via the ear with a tympanic membrane thermometer (Covidiev Genius 2). Systolic and diastolic blood pressure were measured with a calibrated sphygmomanometer from the left arm with the same sphygmomanometer (Erka aneroid sphygmomanometer®) and stethoscope. Pulse rate and respiratory rate were manually monitored for a period of one minute by the researcher using a wristwatch. Verbal and written informed consent was obtained from the subjects or from their closest relatives.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were over 18 years of age and who are able to lie in all positions, and who had unilateral/or bilateral lung disease documented by medical diagnosis by a physician were included in this study.
* Patients who accepted to participated to the study.

Exclusion Criteria:

* Patients who have not accepted to participate.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who were over 18 years of age and who were able to lie in all positions, and who had right lung disease (n=20), left lung disease (n=21) or bilateral lung disease (n=68) documented by medical diagnosis by a physician were included in this descriptive study.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2013-05-12 (Actual); Primary Completion 2013-12-10 (Actual); Study Completion 2015-09-15 (Actual)

PRIMARY OUTCOMES:
oxygen saturation in different positions | an average of 1 year
  SaO2 in each of the five positions

CONTACTS AND LOCATIONS:
Overall Officials: Leyla KHORSHTD, Prof. Dr., Study Director — Ege University

IPD SHARING:
Plan to Share IPD: Yes
The subjects were placed consecutively in random order in the five different positions, SSPB-45°, SSPB-60°, SPB-90°, LRSB-45°, and LLSB-45°, by drawing lots. Oxygen saturation (SaO2) and vital signs (pulse rate, respiratory rate, systolic blood pressure, diastolic blood pressure and body temperature) were measured in each position at 10, 25 and 40 minutes. Oxygen saturation and vital signs were measured with a finger pulse oximeter